CLINICAL TRIAL: NCT06642077
Title: The Effect of Local Anaesthetic Agents on Opioid Use and Recovery in Patients Undergoing Open Heart Surgery: A Randomized Controlled Study
Brief Title: Opioid Use of Local Anaesthetic Agents in Open Heart Surgery and Its Effect on Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hatice AZİZOĞLU, Assist. Prof. Dr., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/19-07
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Analgesics, Opioid; Anesthetics, Local
Keywords: Cardiovascular surgery; Pain management; Local anesthetics; Recovery after surgery; Opioids
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This randomized controlled experimental study was conducted with a total of 60 patients, with 30 patients in the experimental group and 30 patients in the control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): A total of 2 ampoules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml were injected into the sternotomy incision site and around the chest tubes of 30 patients in the experimental group. The total number and dose of opioids, the total number and dose of analgesics used to relieve the pain of the patients in the 24 hours after the injection of 2 ampules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml, and the total number and dose of analgesics were recorded, and the patients were interviewed face-to-face 24 hours later, and Postoperative Recovery Index (PoRI) was recorded.
  Interventions: Drug: LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml
- CONTROL GROUP (No Intervention): No intervention was performed on 30 patients in the control group, and standard treatment and care continued to be applied to these patients.

INTERVENTIONS:
Drug: LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml — A total of 2 ampoules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml were injected into the sternotomy incision site and around the chest tubes of 30 patients in the experimental group. The total number and dose of opioids, the total number and dose of analgesics used to relieve the pain of the patients in the 24 hours after the injection of 2 ampules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml, and the total number and dose of analgesics were recorded, and the patients were interviewed face-to-face 24 hours later, and PoRI was recorded. No intervention was performed on 30 patients in the control group, and standard treatment and care continued to be applied to these patients.
  Other Names: Application of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml to the sternotomy incision area and around the drains
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The aim of this randomized controlled study was to investigate the effect of injecting local anesthetic agents into the sternotomy incision site and around the drains on the amount of opioids used in the postoperative period and the healing process. The main questions it aims to answer are:

* In patients undergoing open heart surgery, does the application of local anesthetic around the sternotomy incision site and chest tube(s) reduce the amount of postoperative opioid use?
* In patients undergoing open heart surgery, does the application of local anesthetic around the sternotomy incision site and chest tube(s) accelerate postoperative recovery?

In this study, LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml will be injected into the sternotomy incision area and around the drains of the patients in the experimental group, and the amount of opioid consumed in the postoperative period will be recorded and the healing process will be observed.

DETAILED DESCRIPTION:
After open heart surgery, patients experience high levels of pain at the sternotomy incision site and around the chest tube(s), affecting their recovery. This study was conducted to determine the effects of local anesthetic application around the sternotomy incision site and chest tube(s) on the amount of opioids used and recovery after surgery in patients undergoing open heart surgery. The study population consisted of patients who underwent open heart surgery in the Cardiovascular Surgery Intensive Care Unit of a hospital. The sample group consisted of patients who met the inclusion criteria (patients between 18 and 65 years of age, conscious, and willing to communicate and cooperate after open heart surgery). For the planned study, the "G. Power-3.1.9.2" program was used to calculate the sample size at an 80% confidence level prior to data collection. The sample was determined with the "Sample Calculation Formula (n=Nz2pq / d2(N-1) + z2pq). According to the literature review, it was determined that the "effect size value was 0.096". Accordingly, with a primary type error of 5% (Z = 1.96), a test power of 80%, and an effect size of 0.096 units, the minimum sample size was calculated as n = 60. Thus, of the 60 volunteer patients included in the study, 30 were randomly assigned to the experimental group and 30 to the control group. Data were collected using a Descriptive Characteristics Form and the Postoperative Recovery Index (PoRI).

A total of 2 ampoules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml were injected into the sternotomy incision site and around the chest tubes of 30 patients in the experimental group. The total number and dose of opioids, the total number and dose of analgesics used to relieve the pain of the patients in the 24 hours after the injection of 2 ampules of LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml, and the total number and dose of analgesics were recorded, and the patients were interviewed face-to-face 24 hours later, and PoRI was recorded. No intervention was performed on 30 patients in the control group, and standard treatment and care continued to be applied to these patients. SPSS 19.0 (SPSS Inc., Chicago, Illinois, USA) package program was used for data evaluation. Descriptive statistics for continuous variables were expressed as mean and standard deviation, while descriptive statistics for categorical variables were expressed as number and percentage. Normality of data distribution was tested by Kolmogorov-Smirnov, and homogeneity of variances was tested by Levene's test. In independent two-group comparisons in terms of continuous variables, the Independent Groups T-test was used in cases where normal distribution conditions were met, and Mann-Whitney U test statistics were used in cases where normal distribution conditions were not met. In independent comparisons of more than two groups in terms of continuous variables, one-way analysis of variance (ANOVA) was used in cases where normal distribution conditions were met, and Kruskal-Wallis test statistics were used in cases where normal distribution conditions were not met. The Spearman rank correlation coefficient was calculated between groups to determine the relationship between continuous variables. All test data were evaluated at a 95% confidence interval and a 0.05 significance level.

Research Hypotheses

H0: In patients undergoing open heart surgery, local anesthetic application around the sternotomy incision site and chest tube(s) has no effect on the amount of postoperative opioid use and recovery.

H1: In patients undergoing open heart surgery, local anesthetic application around the sternotomy incision site and chest tube(s) has an effect on the amount of postoperative opioid use and recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 65 years of age, and willing to communicate and cooperate after open heart surgery

Exclusion Criteria:

* Patients younger than 18 years and older than 65 years, unwilling to communicate and cooperate, sensitive to local anaesthetics and not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Amount of Opioid Consumed in the Postoperative Period | First 24 hours after open heart surgery
  After open heart surgery, LIDOFAST 40 mg/2 ml + 0.025 mg/2 ml will be injected into the sternotomy incision area and around the drains of the patients in the experimental group, and the amount of opioid consumed in the postoperative period will be recorded and compared with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Azizoğlu, Principal Investigator — Yuzuncu Yil University; Mehmet Aşam, Study Chair — Van Training and Research Hospital; Zeynep Gürkan, Study Chair — Yuzuncu Yil University; Yasemin Bozkurt, Study Chair — Van Training and Research Hospital; Canan Demir, Study Chair — Yuzuncu Yil University
Locations (1):
- Yüzüncü Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Ebrahimi S, Paryad E, Ghanbari Khanghah A, Pasdaran A, Kazemnezhad Leili E, Sadeghi Meibodi AM. The effects of lavandula aromatherapy on pain relief after coronary artery bypass graft surgery: A randomized clinical trial. Appl Nurs Res. 2022 Dec;68:151638. doi: 10.1016/j.apnr.2022.151638. Epub 2022 Oct 28. PMID 36473717
- [Result] Choiniere M, Watt-Watson J, Victor JC, Baskett RJ, Bussieres JS, Carrier M, Cogan J, Costello J, Feindel C, Guertin MC, Racine M, Taillefer MC. Prevalence of and risk factors for persistent postoperative nonanginal pain after cardiac surgery: a 2-year prospective multicentre study. CMAJ. 2014 Apr 15;186(7):E213-23. doi: 10.1503/cmaj.131012. Epub 2014 Feb 24. PMID 24566643
- [Result] Cogan J. Pain management after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2010 Sep;14(3):201-4. doi: 10.1177/1089253210378401. PMID 20705642
- [Result] White PF, Rawal S, Latham P, Markowitz S, Issioui T, Chi L, Dellaria S, Shi C, Morse L, Ing C. Use of a continuous local anesthetic infusion for pain management after median sternotomy. Anesthesiology. 2003 Oct;99(4):918-23. doi: 10.1097/00000542-200310000-00026. PMID 14508326
- [Result] Dowling R, Thielmeier K, Ghaly A, Barber D, Boice T, Dine A. Improved pain control after cardiac surgery: results of a randomized, double-blind, clinical trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1271-8. doi: 10.1016/s0022-5223(03)00585-3. PMID 14665996
- [Result] Golembiewski J. Local anesthetics. J Perianesth Nurs. 2013 Dec;28(6):409-12. doi: 10.1016/j.jopan.2013.09.001. No abstract available. PMID 24267631
- [Result] Shah J, Votta-Velis EG, Borgeat A. New local anesthetics. Best Pract Res Clin Anaesthesiol. 2018 Jun;32(2):179-185. doi: 10.1016/j.bpa.2018.06.010. Epub 2018 Jul 3. PMID 30322458
- [Result] Jannati M, Attar A. Analgesia and sedation post-coronary artery bypass graft surgery: a review of the literature. Ther Clin Risk Manag. 2019 Jun 20;15:773-781. doi: 10.2147/TCRM.S195267. eCollection 2019. PMID 31417264
- [Result] Brown CR, Chen Z, Khurshan F, Groeneveld PW, Desai ND. Development of Persistent Opioid Use After Cardiac Surgery. JAMA Cardiol. 2020 Aug 1;5(8):889-896. doi: 10.1001/jamacardio.2020.1445. PMID 32584934
- [Result] Reisli R, Akkaya OT, Arican S, Can OS, Cetingok H, Gulec MS, Koknel Talu G. [Pharmachologic treatment of acute postoperative pain: A clinical practice guideline of The Turkish Society of Algology]. Agri. 2021 Jan;33(Suppl 1):1-51. doi: 10.14744/agri.2021.60243. Turkish. PMID 33523457
- [Derived] Azizoglu H, Asam M, Gurkan Z, Bozkurt Y, Demir C. The effect of local anaesthetic agents on opioid use and recovery in patients undergoing open heart surgery: a randomized controlled study. BMC Cardiovasc Disord. 2025 Feb 1;25(1):72. doi: 10.1186/s12872-025-04493-2. PMID 39893373